CLINICAL TRIAL: NCT02441790
Title: Early Range of Motion in 5th Metacarpal Fracture: A Randomized Controlled Trial
Brief Title: Early Range of Motion in 5th Metacarpal Fracture
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment Difficulty
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIF-2013-07
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Fracture
Keywords: 5th metacarpal; EAROM; standard immobilization; Boxer's Fracture; hand function; DASH; trauma
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Active Range of Motion (Experimental): Early Active Range of Motion (EAROM) 3-9 days following hand fracture
  Interventions: Behavioral: Early Active Range of Motion
- Standard Immoblization (Active Comparator): Standard immobilization with plaster splint for 21-27 following hand fracture
  Interventions: Behavioral: Standard Immobilization

INTERVENTIONS:
Behavioral: Early Active Range of Motion — 3-9 days
  Arms: Early Active Range of Motion
Behavioral: Standard Immobilization — 21-27 days
  Arms: Standard Immoblization

SUMMARY:
Fractures of the fifth metacarpal neck are the most common injury involving the upper extremity. Patients are typically young adult males. Restoring function quickly and reliably for return to work and/or activity is important; these patients are a significant labour force demographic. Treatment is historically splinting for approximately 3-4 weeks. Splinting a fracture is a "trade-off". Immobilization allows stabilization and fracture healing, but also causes hand stiffness and weakness leading to impaired function. Little prospective research exists; there is no agreement for ideal duration of splinting or therapy, demonstrating clinical equipoise. A new concept in hand rehabilitation is "early active range of motion" (EAROM). The objective of this trial is to establish if EAROM provides improved early (6 week) hand function when compared to standard immobilization.

DETAILED DESCRIPTION:
Fractures of the fifth metacarpal neck ("boxer's fractures"), are the most common injury to the upper extremity. They are the result of axial force on a flexed metacarpalphalangeal (MCP) joint. Typically, they are caused by striking a hard object with a closed fist, breaking the knuckle on the "little" finger. Restoring hand function quickly and reliably for return to work and/or activity is of utmost importance. These patients are a significant labour force demographic. Since the injury is not characteristically sustained at work, "return-to-work"is an important patient consideration for lost wages. Treatment for fractures of the fifth metacarpal neck is typically non-operative. In the absence of urgent operative indications (ie. "open fractures" or contamination), non-operative management is initiated. Closed reduction is performed with local anaesthesia and manual manipulation. A splint is then applied. Repeat x-rays are obtained to determine positioning. If anatomic alignment is stable, no surgery is indicated and the patient remains splinted for 3-4 weeks. "Early active range of motion" (EAROM) refers to actively moving the fractured digit once fracture callus has begun formation at 3 days. In practice, EAROM begins at 3-14 days.It involves controlled, active tendon glide exercises where the patient attempts to move joints in the injured hand. This motion is perpendicular to the fractures pattern, applying a compressive force to the fracture. From basic science models, compressive forces of EAROM improve rate of bone callus differentiation,early healing,fracture angulation and load bearing.This study aims to translate these basic science concepts to practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal or greater than 18 years
2. Fifth metacarpal neck fracture, 9 or fewer days since injury
3. Equal or less than 40 degrees of dorsal fracture angulation on lateral x-ray. Angle is measured between the line along the longitudinal axis of the metacarpal shaft and the line from the centre of the metacarpal head to the fracture site.
4. No angulation or malrotation
5. No clinical fracture shortening (ie. Inability to extend fifth digit)
6. Non-operative treatment
7. Volar or ulnar gutter splint (MCP flexed, IPs extended)

Exclusion Criteria:

1. Metabolic bone disease
2. "Open fracture" with soft tissue loss overlying fracture site
3. Tendon injury
4. Neurovascular injury
5. Clinical rotatory malalignment
6. Fracture shortening demonstrated by "pseudoclawing"
7. Other fracture in the ipsilateral upper extremity
8. Any operative indication
9. Previous fracture to the involved fifth ray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Hand function as measured by validated scoring - the Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure | 6 weeks

SECONDARY OUTCOMES:
HR-QOL | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael James Cooper, MD, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada